CLINICAL TRIAL: NCT03267251
Title: Engaging Patients and Providers in Collaborative Communication on HPV Vaccination (EPICC-HPV)
Acronym: EPICC-HPV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Parallel record under the prime awardee (Klein Buendel)
Sponsor: University of New Mexico (Other)
Collaborators: Klein Buendel, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNewMexico
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2017-08

CONDITIONS: Vaccine Decision Making
Keywords: Vaccine Decision Making; Public Health; Health Communication; Digital Interventions

STUDY DESIGN:
Intervention Model Description: This research project will compare usual care clinic-based communication about HPV vaccination (UC) to usual care plus web-based dissemination (UC+GHG) of information on HPV vaccination to parents and adolescent girls using a pair-matched group-randomized pretest-posttest design protocol. Pediatric/family practice clinics in New Mexico (n=30 clinics) will be pair-mated and one clinic per pair will be randomized to UC+GHG condition via the website, GoHealthyGirls.org. The remaining clinic will continue to receive UC only. Assessment protocols will be conducted at pretest, 3-month follow-up, and 9-month follow-up points, measuring knowledge, compatibility and relative advantage principles in DI, shared decision making, and vaccine adoption by girls. Thus, the proposed trial design will be a 2 (UC v. UC+GHG) intervention x 3 (level of time - pretest vs. 3-month follow-up vs. 9-month follow-up) mixed factorial design with participants nested within clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Clinic communication - HPV Vaccine (Active Comparator): Standard Usual and Customary HPV Information - CDC pamphlet
  Interventions: Other: Standard Usual and Customary HPV Information - CDC pamphlet
- Usual Care and Web App on HPV Vaccine (Experimental): Usual Care and Web app on HPV Vaccine: Vacteens Web app for mobile devices
  Interventions: Other: Vacteens Web app for mobile devices

INTERVENTIONS:
Other: Vacteens Web app for mobile devices — The Web app provides parents of young adolescent girls (ages 11-14) accurate information about HPV Vaccination, and a number of tools to aid informed decision making.
  Arms: Usual Care and Web App on HPV Vaccine
Other: Standard Usual and Customary HPV Information - CDC pamphlet — The usual communication about HPV Vaccination in clinics is for parents to be issued the CDC pamphlet on HPV Vaccination.
  Arms: Usual Clinic communication - HPV Vaccine

SUMMARY:
Vaccination against Human Papillomavirus is recommended for adolescent females by the Advisory Committee on Immunization Practices (ACIP), physicians, and many medical organizations, yet uptake of HPV vaccines remains very low. CDC data reveal that in 2013 only 44.3% of 13-17 year old females in New Mexico (and 37.6% nationwide) had completed the 3-dose HPV vaccine series. These data reveal the uptake of the HPV vaccines is unacceptably low, thereby diminishing its ability to provide population-level protection against the HPV types known to cause cervical, vaginal, and vulvar cancers in women, oropharyngeal and anal cancers in men and women, and penile cancers in men. The danger of very low vaccination rates is that adolescents of all ages will continue to be vulnerable to HPV and the associated cancer risks.

Despite recommendations for HPV, parents continue to have concerns about HPV vaccination. Clinicians often lack a clear frame for discussions about HPV vaccination with parents, so much so that recent research indicates that pediatricians' discussions with parents about vaccinations in general often take the form of bargaining, e.g., "since this may be too early for the vaccination, can we delay the vaccination schedule?" Effective messaging is needed to close a knowledge gap among parents around HPV and HPV vaccines, improve communication and shared decision-making about HPV vaccination between adolescent girls' parents and physicians, and ultimately prompt uptake of HPV vaccines.

This project will employ a web-based intervention on HPV as a way to improve knowledge, communication and shared decision-making about HPV vaccination for 11-13 year old girls and their parents. A clinic-based comparative effectiveness randomized trial will be used to examine the impact of the website on vaccine-related outcomes and vaccine uptake. New Mexico pediatric clinics will be randomly assigned to either the usual care clinic-based communication about HPV vaccination or to usual care plus web-based dissemination. Assessments of vaccine-related outcomes, including shared decision-making between girls, parents and physicians, will be assessed at baseline, 3 months, and 9 months and vaccine uptake and dose adherence will be abstracted from clinic vaccine records at 9 months. An effective web-based resource should increase parents' knowledge, intentions and motivations to vaccinate

DETAILED DESCRIPTION:
Uptake of the Human Papillomavirus (HPV) vaccines in the U.S. remains very low. (RQ-1) The quadrivalent HPV vaccine has been routinely recommended for adolescent females by the Advisory Committee on Immunization Practices. The Centers for Disease Control and Prevention (CDC) reports that in 2013, the uptake of HPV vaccines (all three doses) was 37.6% for females (ages 13-17 years). The Healthy People 2020 target for vaccination coverage of adolescent females aged 13-15 years is 80.0% for ≥3 doses of HPV, far above current national rates for HPV vaccine uptake. In New Mexico, the 3-dose completion rate for HPV vaccination for females ages 13-17 is currently 44.3%. However, for girls in the recommended early age vaccination range (11-13), a recent estimate provided by the New Mexico Dept. of Public Health Vaccination Program reveals that in 2012 approximately 7% of 11-12 year old New Mexico adolescent girls completed all 3 doses of HPV vaccine, and in 2013 approximately 9% had completed all 3 doses. In the simplest terms, the uptake of the HPV vaccines is unacceptably low, diminishing its ability to confer population-level protection against the HPV types known to cause cervical, vaginal, and vulvar cancers in women, oropharyngeal and anal cancers in men and women, and penile cancers in men. The danger given the very low vaccination rates reported above is that a significant proportion of adolescents of all ages will not receive the HPV vaccine and continue to be vulnerable to HPV and the associated cancer risks.

Physicians' views of and recommendations for HPV vaccination and parents' perceptions of the HPV vaccines predict HPV vaccine uptake. Despite convincing data on the safety and effectiveness of the vaccines, and a wide variety of medical organizations recommending them, parents continue to have concerns about HPV vaccination. The pattern of vaccine uptake also increases the risk of vaccine-related health disparity across gender and ethnic groups. While minority youth are more likely to begin vaccination programs, they are significantly less likely to complete vaccination programs for reasons that remain in debate. As a result, minority youth lack adequate protection from preventable illnesses. This is particularly problematic as such deficits can build into larger medical consequences later in life.

Diffusion of Innovations theory (DI) provides a framework for explaining vaccine uptake. DI is a theory that seeks to explain how, what, and why new ideas (e.g., vaccines) are spread through different populations at different rates. One tenet of DI is that effective messaging is necessary for the diffusion of a new innovation, and there is a lack of effective messaging to parents to close the knowledge gap about HPV vaccines, resulting in poor uptake. Both the CDC and the President's Cancer Advisory Board call for the development of effective and accessible messaging to improve decision-making around adolescent vaccination, particularly for the HPV vaccines. Effective messaging is especially important to reach minority groups who experience health disparities, especially to parents for whom English may not be the first language. Because parents drive the decision-making around vaccine uptake, messaging should be focused on them, but should include adolescents as well. Clinicians also often lack a clear frame for discussions about HPV vaccination with parents. The topic of vaccines is a polarizing one for many physicians and their patients (parents and children). Physicians often find their expertise and recommendations being accepted by parents for certain areas of their child's care (e.g., diet, seatbelt use), but not others. Providers are using many strategies in response, but think few are effective. Very little research has been conducted on clinic interventions that improve vaccine uptake, or on interventions that would help physicians effectively frame HPV vaccination discussion with parents. With the recent approval of the new 9-valent vaccine (Gardasil 9), a further premium is placed on effective communication between parents and physicians communicating about HPV vaccines. The focus in this project is to employ a developed and efficacious digital intervention on HPV messaging (GoHealthyGirls.org) as a way to improve the communication and shared decision-making about HPV vaccination between girls' parents and pediatricians. An effective web-based resource in pediatric and family practice clinics should increase parents' knowledge, intentions and motivations to vaccinate, enhance pediatrician-parent shared decision making for HPV vaccination, and increase HPV vaccination rates.

A clinic-based comparative effectiveness randomized trial will be used to examine the impact of the GoHealthyGirls website on vaccine-related outcomes and vaccine uptake. Pediatric clinics within established health care networks in New Mexico will be randomly assigned to either the usual care clinic-based communication about HPV vaccination (UC) or to usual care plus web-based dissemination (UC+GHG). Assessments of vaccine-related outcomes, including shared decision making between parents and physicians, will be assessed at baseline, 3 months, and 9 months. Vaccine uptake and dose adherence will be abstracted from clinic vaccine records. Comparative effectiveness, sensitivity analysis, and heterogeneity of treatment effects analyses are planned. An extensive parent and stakeholder engagement plan will be utilized, and includes an Adolescent HPV Immunization Advocacy Coalition that will involve parents across New Mexico, and an Adolescent HPV Immunization Expert Advisory Board that will involve clinicians, vaccine experts and researchers in New Mexico. Quarterly meetings of these groups will review project plans, protocols, and processes, and link the project to the communities and population of New Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Parent of an adolescent girl ages 11-14, adolescent girl has not yet received HPV vaccination

Exclusion Criteria:

* adolescent girl has received HPV vaccination

Min Age: 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Vaccine Adoption | 9-month follow up
  Shot records of initial and second HPV vaccination

SECONDARY OUTCOMES:
Parental HPV vaccination knowledge - questionnaire | Baseline, 3-month and 9-month follow-up
  Assessment of HPV-related knowledge among parents, developed by Perez, et al.
Shared decision-making (SDM-Q9) questionnaire | 3-month and 9-month follow-up
  Assessment of Shared Decision Making, developed by Kriston, et al.
Physician-Patient Communication questionnaire | 3-month and 9-month follow-up
  Satisfaction of communication between healthcare provider and parent, developed by Street, et al.

CONTACTS AND LOCATIONS:
Overall Officials: William Lawrence, MD, Study Chair — Patient Centered Outcomes Research Organization

IPD SHARING:
Plan to Share IPD: No
No plan at this time.